CLINICAL TRIAL: NCT05000697
Title: Chemoradiation and Consolidation Chemotherapy With or Without Oxaliplatin for Distal Rectal Cancer and Watch and Wait. A Multi-center Prospective Randomized Controlled Trial. (CCHOWW)
Brief Title: Chemoradiation and Consolidation Chemotherapy With or Without Oxaliplatin for Distal Rectal Cancer and Watch and Wait
Acronym: CCHOWW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Alemão Oswaldo Cruz (Other)
Responsible Party: Principal Investigator, Rodrigo Oliva Perez, Principal Investigator, Hospital Alemão Oswaldo Cruz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 46102621.3.1001.0070
Record Dates: First submitted 2021-07-19; First posted 2021-08-11 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Rectal Cancer; Consolidation
Keywords: Rectal cancer; Consolidation Chemotherapy; Complete Response; Watch and Wait
MeSH Terms: conditions — Rectal Neoplasms; Pathologic Complete Response | interventions — Oxaliplatin; Fluorouracil

STUDY DESIGN:
Intervention Model Description: Individuals will be randomized and allocated at a 1:1 ratio to the two groups using a permuted block design with a random block size of 4, 6, and 8. (1-3) A randomization list will be generated electronically using appropriate software immediately after being considered eligible.
Who Masked: Investigator
Masking Description: Patients and attending phisicians will not be blinded to the treatment arm randomized for each patient. However, as a strategy to reduce investigator's expectations and reduce inherent bias, the central committee will be blinded to the treatment arm. It is expected that blinding the central committee, who will be responsible for assessing the primary endpoint, any bias related to the investigator's expectation about the treatment arm and the chances of Watch and Wait will be nulled.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 - 5FU + Oxaliplatin (Experimental): 1) RT (54Gy) plus daily concomitant capecitabine 825mg/m2 bid, followed by mFOLFOX6 or XELOX for 4 cycles (12 weeks), starting 1 week after radiotherapy ended;
  Interventions: Drug: Oxaliplatin; Drug: 5FU
- Arm 2 - 5FU Only (Active Comparator): 2) RT (54Gy) plus daily concomitant capecitabine 825mg/m2 bid, followed by capecitabine 2000mg/m2/day for 14 days in a 21 days cycle for 4 cycles (12 weeks), starting 1 week after radiotherapy ended;
  Interventions: Drug: 5FU

INTERVENTIONS:
Drug: Oxaliplatin — Patients will receive 5FU + Oxaliplatin during the consolidation chemotherapy after long course chemoradiation
  Other Names: 5FU + Oxaliplatin
  Arms: Arm 1 - 5FU + Oxaliplatin
Drug: 5FU — Patients will receive 5FU during the consolidation chemotherapy after long course chemoradiation

SUMMARY:
Background: Neoadjuvant chemoradiation (nCRT) has been considered the preferred initial treatment strategy for distal rectal cancer. Advantages of this approach include improved local control after radical surgery but also the opportunity for organ preserving strategies (Watch and Wait - WW). Consolidation chemotherapy (cCT) regimens using fluoropyrimidine-based with or without oxaliplatin following nCRT have demonstrated to increase complete response and organ preservation rates among these patients. However, the benefit of adding oxaliplatin to cCt compared to fluoropyrimidine alone regimens in terms of primary tumor response remains unclear. Since oxaliplatin-treatment may be associated with considerable toxicity, it becomes imperative to understand the benefit of its incorporation into standard cCT regimens in terms of primary tumor response. The aim of the present trial is to compare the outcomes of 2 different cCT regimens following nCRT (fluoropyrimidine-alone versus fluoropyrimidine+oxaliplatin) for patients with distal rectal cancer.

Methods: In this multi-centre study, patients with magnetic resonance-defined distal rectal tumors will be randomized on a 1:1 ratio to receive long-course chemoradiation (54Gy) followed by cCT with fluoropyrimidine alone versus fluoropyrimidine+oxaliplatin. Magnetic resonance (MR) will be analyzed centrally prior to patient inclusion and randomization. mrT2-3N0-1 tumor located no more than 1cm above the anorectal ring determined by sagittal views on MR will be eligible for the study. Tumor response will be assessed after 12 weeks from radiotherapy (RT) completion. Patients with clinical complete response (clinical, endoscopic and radiological) will be enrolled in an organ-preservation program (WW). The primary endpoint of this trial is decision to organ-preservation surveillance (WW) at 18 weeks from RT completion.

Discussion: Long-course nCRT with cCT is associated with improved complete response rates and may be a very attractive alternative to increase the chances for organ-preservation strategies. Fluoropyrimidine-based cCT with or without oxaliplatin has never been investigated in the setting of a randomized trial to compare clinical response rates and the possibility of organ-preservation. The outcomes of this study may significantly impact clinical practice of patients with distal rectal cancer interested in organ-preservation.

DETAILED DESCRIPTION:
Patients and Methods

Patients with distal rectal cancer will be eligible for the study after initial clinical, endoscopic and radiological assessment. At this point, patients will be offered to participate in the study and after informed consent, randomized to control or experimental arms as follows.

Endpoints

Primary endpoint: Decision to Watch and Wait due to clinical complete response achieved at 18 weeks from last date of radiation using clinical (DRE), endoscopic and radiological criteria (mrTRG grade) or near-complete clinical response (no progressive disease clinically, endoscopically or radiologically)

Definition of clinical complete response (cCR) available below and at the discretion of the attending surgeon.

Definition of radiological complete response as described below (centralized).

Patients will be counted as event if at 18 weeks the decision is to interrupt Watch and Wait and proceed to surgery (any kind) because of overt incomplete clinical response. In order to standardize assessment of response and reduce inter-observer variability, the decision to continue on Watch and Wait (or not) will be at the discretion of the central committee during central revision of studies.

Secondary endpoints:

* Surgery-free survival at 3 years
* TME-free survival at 3 years
* Distant metastases free survival at 3 years
* Local regrowth-free survival at 3 years
* Colostomy-free survival at 3 years

Definitions

Definition of cCR:

* Endoscopic: white scar, teleangiectasia, absence of ulceration and/or mass 6
* Clinical: no irregularity, firm area with minor induration6
* Radiological: mrTRG1: fibrosis with low signal intensity seen on T2 weighted images replacing the primary tumor; no restricted diffusion on diffusion weighted images; no nodes with border irregularity or mixed signal intensity; no extramural vascular invasion23-26

Definition of near-complete response:

* Endoscopic: residual tumor size ≤2cm (or reduction of ≥70% original tumor volume/size) 4,27,28
* Clinical: only superficial ulceration or minor (questionable) irregularities of the mucosal/rectal wall
* Radiological: mrTRG2 predominant fibrosis with low signal with foci of intermediate tumor signal intensity seen on T2 weighted images with or without restricted diffusion; mrTRG1: fibrosis with low signal intensity seen on T2 weighted images replacing the primary tumor with restricted diffusion; no nodes with border irregularity or mixed signal intensity; no extramural vascular invasion 27

Central Committee

The central committee is multidisciplinary group of surgeons, medical oncologists and radiologists previously appointed at the beginning of the recruitment of patients and with previous experience with organ preservation.2, 21 This group of specialist will be responsible to assess the baseline staging and define if the patients fulfill all the inclusion/exclusion criteria prior to randomization. The committee will also be responsible to evaluate the endoscopic and radiological tumor re-assessment studies at 12 and 18 weeks from radiation completion. The definition to continue on the Watch and Wait pathway or not will be at the discretion of this committee.

Technical aspects of assessment tests:

Suggested MR protocol:

1.5T - FRFSE; TR/TE: 3300/120 (ms); slice thickness/gap: 3.0/0; Matrix: 256 x 256; NSA 8) 3.0T - FRFSE; TR/TE: 8000/150 (ms); slice thickness/gap: 3.0/0; Matrix: 288 x 288; NSA 5) DWI - inclusion of a high b-value of at least 800

Suggested Endoscopic assessment:

Endoscopic assessment using a flexible scope (gastroscope preferred for retroflexion); direct endoscopic and retroflexion view of the primary tumor/scar; endoscopic biopsies at discretion of participating center.

Radiotherapy

Preoperative radiotherapy will be delivered on a linear accelerator in prone or supine position, preferably with full bladder. The use of a belly board is allowed. Isocentric 3 or 4 fields, as well as an IMRT technique is allowed, as long as all beams are treated on a daily basis. The dose distribution and calculation should be performed on CT or MRI and specified according to the ICRU 50 guidelines.

Dose specification: All patients will receive 25 daily fractions of 1.8 Gy up to a total dose of 45 Gy to the pelvic field including the tumor bed with a margin and the regional lymph nodes. A field reduction after 45 Gy is recommended up to 54 Gy. The last 5 fractions will then be given to the tumor bed with a margin.

Target volume:

Pelvic CTV

* The primary tumor
* Mesorectum: Distally, only lymph nodes or tumor deposits up to 4 cm are included. For tumors in lower rectum this means that the entire mesorectum down to the pelvic floor is included.
* Presacral nodes and nodes along the rectal superior artery: Since local recurrences are very unusual above S1 - S2, lymph nodes above this level should not be included unless there are signs of radiologically positive lymph nodes presacrally. If this is the case, the cranial limit of CTV should be at least 1 cm above the most cranial radiologically positive lymph node.
* Lateral lymph node stations: Until they reach the level of the obturator canal Internal iliac artery up to the bifurcation from the external iliac artery. The cranial border for the CTV is in most cases just below the bifurcation of the internal and external iliac arteries. In most patients this is at the level of S1 - S2.
* Ischio-rectal fossa and the anal canal: Included in pelvic CTV only if the tumor grows into the levators or down into the anal canal.
* Lymph nodes along the external iliac artery: Included if the tumor grows into anterior organs like the prostate, urinary bladder, cervix, vagina or uterus to such an extent that the external nodes are at risk for metastases.

Boost GTV:

GTV is the visible primary tumor and radiologically positive lymph nodes.

CTV boost:

GTV boost plus a margin of 2 cm within the same anatomical compartment as the tumour is in, for the dose of 45 Gy, also around radiologically engaged lymph nodes.

PTV:

The above description relates to the CTV. A PTV should normally be defined and includes CTV and internal target volume (ITV) and a margin necessary for the setup. These margins are depending upon several factors that are related to the equipment at each radiotherapy center.

Chemotherapy Protocols

Concomitant chemotherapy:

Concomitant capecitabine: 825mg/m2 bid on the radiotherapy days only

Consolidation chemotherapy:

1. Consolidation capecitabine (alone): 1000mg/m2 bid, for 14 days, in a 3 week cycle, for 4 cycles
2. Consolidation options with oxaliplatin:

2.1. mFOLFOX6: Oxaliplatin 85mg/m2 plus Leucovorin 400mg/m2 on a concomitant 2 hours infusion. 5FU 400mg/m2 on a bolus infusion, followed by 5FU 2400mg/m2 in 46 hours infusion, every 2 weeks, for 6 cycles 2.2. CAPOX: Oxaliplatin 130mg/m2 on a 2 hours infusion. Capecitabine 1000mg/m2 bid daily, for 14 days, starting on the evening of the oxaliplatin infusion. Repeat every 3 weeks, for 4 cycles

Assessment of Response

Assessment of response will be performed at 12 weeks (and 18 weeks from last date of radiation therapy if cCR or near-complete response is detected at 12 weeks). All patients will undergo endoscopic reassessment, DRE and high-resolution MR. Endoscopic biopsies will be at the discretion of the attending surgeon/endoscopist.

Patients with complete or near-complete clinical response at 12 weeks will be recommended reassessment at 18 weeks from RT. Patients with clinically overt incomplete clinical response at 12 or 18 weeks will be referred to immediate radical surgery.

Randomization

Individuals will be randomized and allocated at a 1:1 ratio to the two groups (control and experimental) using a permuted block design with a random block size of 4, 6, and 8. (1-3) A randomization list will be generated electronically using appropriate software immediately after being considered eligible.

Protocol Blinding

Patients and attending physicians will not be blinded to the treatment arm randomized for each patient. However, as a strategy to reduce investigator's expectations and reduce inherent bias, the central committee will be blinded to the treatment arm. It is expected that blinding the central committee, who will be responsible for assessing the primary endpoint, any bias related to the investigator's expectation about the treatment arm and the chances of Watch and Wait will be nulled.

Sample size calculation

The primary endpoint (decision to WW due to cCR/near CR) was observed in 55% and 85% at 12 weeks (in contrast to the 18 weeks used in the present trial) among patients with early cT3 and cT2 rectal cancer respectively.29 In this study, there was a distribution of 66% of cT3 and 33% cT2. Therefore, response rates appear to be highly dependent on exact T-stage distribution. Considering the expected inclusion of more advanced disease (late mrT3 or even mrT4 rectal cancers) the investigators expect 40% cCR/near-CR in the control arm. A similar difference 60% versus 40% was achieved in the preliminary report of the outcomes of the OPRA trial. This difference in TME-free survival at 3 years was statistically significant favoring patients undergoing nCRT with cCT in comparison to nCRT preceded by induction chemotherapy (both regimens incorporating oxaliplatin). In this setting, if experimental results in ≥60% cCR/near-CR, the study will be considered POSITIVE. The incorporation of oxaliplatin to a consolidation CRT regimen that results in ≥20% increase in cCR/near-CR exceeds the potential disadvantages of treatment-related toxicity.

The investigators will assume that the primary outcome will occur in 40% of individuals in control group and 60% in the experimental group, which corresponds to an absolute difference in proportions of 20%. It is estimated that a sample of 194 (97 per group) provides 80% statistical power to detect this difference at a significance level of 5% using the Chi-square test and assuming a two-sided significance hypothesis and considering a 1:1 allocation. The estimated dropout rate is 10% in each group, so it is expected to include 216 individuals (108 per group). The sample size calculation was performed using SAS 9.4 (PROC POWER procedure).

Time-table

Patient accrual: 2 years and 6 months Patient/institution/year: 5-6 (20 institutions: 100-120/year - 2 years n=200-240)

Interim analysis:

If the arm of two drugs during consolidation shows ≥25% response rate after 72 patients, study will be interrupted (efficacy). If the arm of two drugs shows less than 5% response rate after 72 patients, the study will be interrupted.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. ECOG 0-2 or KPS≥70;
3. Primary rectal adenocarcinoma (biopsy confirmed) within the reach of digital rectal examination (at least lower tip/border) by the attending colorectal surgeon;
4. Endoscopic documentation;
5. Abdominal and chest CT scans showing no evidence of metastatic disease;
6. High-resolution magnetic resonance images performed at either 1.5T or 3.0T system using a phased array surface coil with: sagittal T2 images including the anal verge and the sacrum; axial oblique T2 weighted images acquired in a plane perpendicular to the long axis of the rectal wall guided by the sagittal images; coronal images acquired in parallel to the anal canal plane. Small field of view (16-18cm), 3mm section thickness, increased matrix size and increased number of signal averages are required;
7. Radiological defining criteria (centralized):

   1. Lower edge of tumor at the level (max. 1cm distance) or below the anorectal ring defined at sagittal or coronal views;
   2. mrT2, mrT3 (any subclassification)
   3. mrN0-1 (≤3 radiologically positive lymph nodes)
   4. mrEMVI: any status
   5. mrMRF: any status

Exclusion Criteria:

1. Pregnancy
2. ECOG ≥3 or KPS<70
3. Unwilling to consent
4. Metastatic disease (any kind; internal iliac and obturator nodes are considered local disease and not metastatic disease and therefore will not be considered as exclusion criteria)
5. mrT4 or mrN2
6. Previous pelvic irradiation
7. Baseline neuropathy
8. Receiving treatment of other anti-cancer drug or methods
9. Presence of uncontrolled life threatening diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Decision to Watch and Wait due to clinical complete response | 18 weeks from last date of radiation
  Decision to Watch and Wait due to clinical complete response achieved at 18 weeks from last date of radiation using clinical (DRE), endoscopic and radiological criteria (mrTRG grade) or near-complete clinical response (no progressive disease clinically, endoscopically or radiologically)

SECONDARY OUTCOMES:
Surgery-free survival at 3 years | 3 years from last date of radiation
  Investigate the risk of being surgery-free after 3 years from radiation completion according to the treatment arm
Total Mesorectal Excision-free survival at 3 years | 3 years from last date of radiation
  Investigate the risk of being total mesorectal excision-free after 3 years from radiation completion according to the treatment arm
Distant metastases free survival at 3 years | 3 years from last date of radiation
  Investigate the risk of being distant metastases-free after 3 years from radiation completion according to the treatment arm
Local regrowth-free survival at 3 years | 3 years from last date of radiation
  Investigate the risk of being local regrowth-free after 3 years from radiation completion according to the treatment arm
Colostomy-free survival at 3 years | 3 years from last date of radiation
  Investigate the risk of being colostomy-free after 3 years from radiation completion according to the treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo O Perez, Dr, Principal Investigator — Hospital Alemão Oswaldo Cruz
Locations (24):
- Argentina (5):
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Ramos Mejia: Hospital General de Agudos Dr. Jose Maria Ramos Mejia, Buenos Aires
  - Hospital de Gastroenterologia Udaondo Ciudad de Buenos Aires, Buenos Aires
  - Hospital Britanico de Buenos Aires - Asociacion Civil, Buenos Aires
  - Hospital Curruca: Superintendencia de Bienestar Policia Federal Argentina, Buenos Aires
- Brazil (18):
  - Hospital Alemão Oswaldo Cruz, São Paulo, São Paulo
  - Hospital Felicio Rocho, Belo Horizonte
  - Hospital das Clínicas da Faculdade de Medicina de Botucatu, Botucatu
  - Complexo de Saude São João de Deus - Divinopolis, Divinópolis
  - Hospital das Clinicas de Passo Fundo, Passo Fundo
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - União Brasileira de Educação e Assistencia - PUC-RS - Campus POA, Porto Alegre
  - Hospital Militar de Area de Porto Alegre, Porto Alegre
  - Centro Gaucho Integrado de Oncologia, hematologia, ensino e pesquisa, Porto Alegre
  - Instituto Nacional do Cancer Jose Alencar Gomes da Silva - INCA, Rio de Janeiro
  - Ensino e Terapia de Inovação Clínica AMO, Salvador
  - Hospital Universitário de Santa Maria, Santa Maria
  - Hospital Beneficencia Portuguesa, São Paulo
  - Associação Beneficente Síria - Hospital do Coração, São Paulo
  - Centro Paulista de Oncologia - CPO, São Paulo
  - Hospital Primavera, São Paulo
  - COT - Centro Oncológico do Triângulo S.A., Uberlândia
- Médica Uruguaya Coorporación de Asistencia Médica, Montevideo, Uruguay

REFERENCES:
- [Derived] Habr-Gama A, Sao Juliao GP, Ortega CD, Vailati BB, Araujo S, Jorge T, Sabbaga J, Rossi GL, D'Alpino R, Kater FR, Aguilar PB, Mattacheo A, Perez RO; Latin American Rectal Cancer Consortium (LARCC). A multi-centre randomized controlled trial investigating Consolidation Chemotherapy with and without oxaliplatin in distal rectal cancer and Watch & Wait. BMC Cancer. 2023 Jun 14;23(1):546. doi: 10.1186/s12885-023-10984-2. PMID 37316784

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Statistical Analysis Plan (2024-01-23): https://cdn.clinicaltrials.gov/large-docs/97/NCT05000697/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT05000697/ICF_002.pdf